CLINICAL TRIAL: NCT04047004
Title: Adjuvant Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) During Laparoscopic Resection in High-risk Gastric Cancer Patients: A Multicentre Phase-I Study (the PIPAC-OPC4 Study)
Brief Title: Adjuvant PIPAC in Gastric Cancer Patients
Acronym: PIPAC-OPC4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Michael Bau Mortensen (Other)
Responsible Party: Sponsor-Investigator, Michael Bau Mortensen, Professor, Consultant, DMSci, PhD, MD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PIPAC-OPC4
Record Dates: First submitted 2019-08-02; First posted 2019-08-06 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Gastric Adenocarcinoma; Gastric Cancer
Keywords: Gastric adenocarcinoma; Intraperitoneal chemotherapy; Laparoscopic gastrectomy; Gastric cancer; Surgery
MeSH Terms: conditions — Stomach Neoplasms | interventions — Doxorubicin; Cisplatin

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, non-randomized, non-blinded, open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-risk gastric cancer patients (Experimental): The study population of high-risk gastric cancer patients will be offered one session of PIPAC immediately after laparoscopic removal of the stomach.
  Interventions: Drug: Doxorubicin; Drug: Cisplatin

INTERVENTIONS:
Drug: Doxorubicin — Conventional PIPAC with doxorubicin (2.1 mg/m2 body surface in 50ml saline) is performed through the CE-certified nebulizer by certified PIPAC surgeons directly after the completion of the laparoscopic gastric resection and reconstruction using the remaining relevant ports. Chemotherapy is installed at a rate of 0.5-0.8 ml/s with a maximum pressure of 300 pressure per square inch and 30 minutes of simple diffusion.
Drug: Cisplatin — Conventional PIPAC with cisplatin (10.5 mg/m2 body surface in 150ml saline) is performed through the CE-certified nebulizer by certified PIPAC surgeons directly after the completion of the laparoscopic gastric resection and reconstruction using the remaining relevant ports. Chemotherapy is installed at a rate of 0.5-0.8 ml/s with a maximum pressure of 300 pressure per square inch and 30 minutes of simple diffusion.

SUMMARY:
In this study patients will be offered intraperitoneal atomized chemotherapy as a supplement to the standard treatment of high-risk gastric cancer (laparoscopic removal of the stomach). Two commercially available oncologic drugs will be used (doxorubicin and cisplatin).

DETAILED DESCRIPTION:
Gastric adenocarcinoma (GAC) is considered the fifth most common cancer in the word and the third leading cause of cancer death globally. The majority of GAC patients presents with advanced stages of disease leading to a dismal prognosis even after treatments with curative intent.

Irrespective of these tumors' origin, the peritoneum is one of the most frequent sites of metastases and recurrences that generally determines the subsequent prognosis. Additionally, it is observed that none of the currently available perioperative chemotherapy regimens have been able to reduce the risk for peritoneal deposits. Peritoneal metastases (PMs) are formed during processes that entraps the malignant cells and this restrictive milieu is thought to hinder the penetrance of drugs delivered systemically and provides grounds for the early administration of intraperitoneal treatments. The presence of malignant intraperitoneal cells that is not cleared by chemotherapy before surgery, and/or seeding of malignant cells during surgery, are probably the major reasons for the development of PM and thus the poor prognosis after seemingly micro-radical surgery.

Since only a fraction of the systemically administered chemotherapy reaches the peritoneum, the effect of intraperitoneal chemotherapy has been eagerly studied. A recent systematic review and meta-analysis identified three trials evaluating the effect of intraperitoneal chemotherapy and/or extensive peritoneal lavage in gastric cancer patients who underwent subsequent surgery. Two and five-year overall survival increased significantly in patients who had intraperitoneal chemotherapy (RR=1.62 and 3.10) and survival further increased by the addition of extensive lavage (RR= 2.33 and 6.19).

The intraperitoneal delivery and subsequent uptake of chemotherapy is improved by a new aerosol technique. Pressurized Intraperitoneal Aerosol Chemotherapy (PIPAC) has shown promising results in patients with PM from colorectal, ovarian and gastric cancer (see below), and PIPAC is feasible, safe and well tolerated by the majority of patients. Our own database assessed the outcome of PIPAC, with low-dose cisplatin and doxorubicin, in GAC patients with chemotherapy-resistant PM. Objective tumor response was documented in 40% of the patients after PIPAC, including complete histological regression in some, whereas an additional 20% had no further tumor progression (manuscript in preparation). These observations in GAC patients deliver further evidence suggesting that PIPAC can induce regression of resistant PMs in several cancer types and might meet the clinical need for new and better therapies for fatal cancer disease states. Our results also provide evidence that low-dose PIPAC therapy might be effective in treating patients with recurrent, chemo-resistant gastric PMs, including the aggressive signet-ring histology.

The imminent question is whether PIPAC delivered immediately after a laparoscopic gastrectomy for GAC, in patients being exposed to a significant risk of early recurrent disease, can be safely carried out? If so, for the first time, a corresponding therapeutic concept can be offered to similar GAC patients in addition to surgery with curative intent. This could potentially increase progression free and eventually overall survival.

Twenty patients will be enrolled from two Danish and Swedish hospitals according to the inclusion and exclusion criteria and included in the data analysis if laparoscopic removal of the stomach and subsequent immediate PIPAC has been performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with high-risk GAC defined as: Diffuse cancer (signet ring cells predominant) or clinical stage: cTany + cN2-3 or cT3-T4 + cNany or GAC patients with preoperative positive peritoneal cytology submitted to laparoscopic gastrectomy (+/- neoadjuvant treatment).
* Age 18 or above
* Written informed consent
* Women must be postmenopausal or use adequate contraception with a negative pregnancy test at inclusion.

Exclusion Criteria:

* Previous allergic reaction to cisplatin, doxorubicin or other platinum containing compounds.
* Renal impairment, defined as GFR < 40 ml/min (Cockcroft-Gault Equation).
* Myocardial insufficiency, defined as NYHA class 3-4.
* Impaired liver function defined as bilirubin ≥ 1.5 x UNL (upper normal limit).
* Inadequate haematological function defined as absolute neutrophil count (ANC) ≤ 1.5 x 10^9/l and platelets ≤ 100 x 10^9/l.
* Any other condition or therapy, which in the investigator's opinion may pose a risk to the patient or interfere with the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Medical adverse events | 30 days
  According to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.
Surgical complications | 30 days
  According to the Dindo-Clavien classification

SECONDARY OUTCOMES:
Length of stay | 30 days
  The amount of time the patient is hospitalized
Positive peritoneal lavage | 30 days
  The rate of positive peritoneal lavage before and after surgery
Adjuvant chemotherapy | 30 days
  The number of patients that receive adjuvant systemic chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Signe Bremholm Ellebæk, MD, PhD, Principal Investigator — Odense University Hospital
Locations (2):
- Odense PIPAC Center, Department of Surgery, Odense University Hospital, Odense, Denmark
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yang D, Hendifar A, Lenz C, Togawa K, Lenz F, Lurje G, Pohl A, Winder T, Ning Y, Groshen S, Lenz HJ. Survival of metastatic gastric cancer: Significance of age, sex and race/ethnicity. J Gastrointest Oncol. 2011 Jun;2(2):77-84. doi: 10.3978/j.issn.2078-6891.2010.025. PMID 22811834
- [Background] Wagner AD, Syn NL, Moehler M, Grothe W, Yong WP, Tai BC, Ho J, Unverzagt S. Chemotherapy for advanced gastric cancer. Cochrane Database Syst Rev. 2017 Aug 29;8(8):CD004064. doi: 10.1002/14651858.CD004064.pub4. PMID 28850174
- [Background] Al-Batran SE, Homann N, Pauligk C, Illerhaus G, Martens UM, Stoehlmacher J, Schmalenberg H, Luley KB, Prasnikar N, Egger M, Probst S, Messmann H, Moehler M, Fischbach W, Hartmann JT, Mayer F, Hoffkes HG, Koenigsmann M, Arnold D, Kraus TW, Grimm K, Berkhoff S, Post S, Jager E, Bechstein W, Ronellenfitsch U, Monig S, Hofheinz RD. Effect of Neoadjuvant Chemotherapy Followed by Surgical Resection on Survival in Patients With Limited Metastatic Gastric or Gastroesophageal Junction Cancer: The AIO-FLOT3 Trial. JAMA Oncol. 2017 Sep 1;3(9):1237-1244. doi: 10.1001/jamaoncol.2017.0515. PMID 28448662
- [Background] Al-Batran SE, Hofheinz RD, Pauligk C, Kopp HG, Haag GM, Luley KB, Meiler J, Homann N, Lorenzen S, Schmalenberg H, Probst S, Koenigsmann M, Egger M, Prasnikar N, Caca K, Trojan J, Martens UM, Block A, Fischbach W, Mahlberg R, Clemens M, Illerhaus G, Zirlik K, Behringer DM, Schmiegel W, Pohl M, Heike M, Ronellenfitsch U, Schuler M, Bechstein WO, Konigsrainer A, Gaiser T, Schirmacher P, Hozaeel W, Reichart A, Goetze TO, Sievert M, Jager E, Monig S, Tannapfel A. Histopathological regression after neoadjuvant docetaxel, oxaliplatin, fluorouracil, and leucovorin versus epirubicin, cisplatin, and fluorouracil or capecitabine in patients with resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4-AIO): results from the phase 2 part of a multicentre, open-label, randomised phase 2/3 trial. Lancet Oncol. 2016 Dec;17(12):1697-1708. doi: 10.1016/S1470-2045(16)30531-9. Epub 2016 Oct 22. PMID 27776843
- [Background] Cunningham D, Allum WH, Stenning SP, Thompson JN, Van de Velde CJ, Nicolson M, Scarffe JH, Lofts FJ, Falk SJ, Iveson TJ, Smith DB, Langley RE, Verma M, Weeden S, Chua YJ, MAGIC Trial Participants. Perioperative chemotherapy versus surgery alone for resectable gastroesophageal cancer. N Engl J Med. 2006 Jul 6;355(1):11-20. doi: 10.1056/NEJMoa055531. PMID 16822992
- [Background] Bringeland EA, Wasmuth HH, Gronbech JE. Perioperative chemotherapy for resectable gastric cancer - what is the evidence? Scand J Gastroenterol. 2017 Jun-Jul;52(6-7):647-653. doi: 10.1080/00365521.2017.1293727. Epub 2017 Feb 28. PMID 28276825
- [Background] Takebayashi K, Murata S, Yamamoto H, Ishida M, Yamaguchi T, Kojima M, Shimizu T, Shiomi H, Sonoda H, Naka S, Mekata E, Okabe H, Tani T. Surgery-induced peritoneal cancer cells in patients who have undergone curative gastrectomy for gastric cancer. Ann Surg Oncol. 2014 Jun;21(6):1991-7. doi: 10.1245/s10434-014-3525-9. Epub 2014 Feb 6. PMID 24499832
- [Background] De Andrade JP, Mezhir JJ. The critical role of peritoneal cytology in the staging of gastric cancer: an evidence-based review. J Surg Oncol. 2014 Sep;110(3):291-7. doi: 10.1002/jso.23632. Epub 2014 May 22. PMID 24850538
- [Background] Minchinton AI, Tannock IF. Drug penetration in solid tumours. Nat Rev Cancer. 2006 Aug;6(8):583-92. doi: 10.1038/nrc1893. PMID 16862189
- [Background] Bentrem D, Wilton A, Mazumdar M, Brennan M, Coit D. The value of peritoneal cytology as a preoperative predictor in patients with gastric carcinoma undergoing a curative resection. Ann Surg Oncol. 2005 May;12(5):347-53. doi: 10.1245/ASO.2005.03.065. Epub 2005 Mar 31. PMID 15915368
- [Background] Ji ZH, Peng KW, Li Y. Intraperitoneal free cancer cells in gastric cancer: pathology of peritoneal carcinomatosis and rationale for intraperitoneal chemotherapy/hyperthermic intraperitoneal chemotherapy in gastric cancer. Transl Gastroenterol Hepatol. 2016 Sep 19;1:69. doi: 10.21037/tgh.2016.08.03. eCollection 2016. PMID 28138635
- [Background] Coccolini F, Catena F, Glehen O, Yonemura Y, Sugarbaker PH, Piso P, Ceresoli M, Montori G, Ansaloni L. Effect of intraperitoneal chemotherapy and peritoneal lavage in positive peritoneal cytology in gastric cancer. Systematic review and meta-analysis. Eur J Surg Oncol. 2016 Sep;42(9):1261-7. doi: 10.1016/j.ejso.2016.03.035. Epub 2016 Apr 19. PMID 27134147
- [Background] Grass F, Vuagniaux A, Teixeira-Farinha H, Lehmann K, Demartines N, Hubner M. Systematic review of pressurized intraperitoneal aerosol chemotherapy for the treatment of advanced peritoneal carcinomatosis. Br J Surg. 2017 May;104(6):669-678. doi: 10.1002/bjs.10521. PMID 28407227
- [Background] Graversen M, Lundell L, Fristrup C, Pfeiffer P, Mortensen MB. Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC) as an outpatient procedure. Pleura Peritoneum. 2018 Nov 27;3(4):20180128. doi: 10.1515/pp-2018-0128. eCollection 2018 Dec 1. PMID 30911669
- [Background] Graversen M, Detlefsen S, Bjerregaard JK, Fristrup CW, Pfeiffer P, Mortensen MB. Prospective, single-center implementation and response evaluation of pressurized intraperitoneal aerosol chemotherapy (PIPAC) for peritoneal metastasis. Ther Adv Med Oncol. 2018 Jun 1;10:1758835918777036. doi: 10.1177/1758835918777036. eCollection 2018. PMID 29899763
- [Background] Graversen M, Pedersen PB, Mortensen MB. Environmental safety during the administration of Pressurized IntraPeritoneal Aerosol Chemotherapy (PIPAC). Pleura Peritoneum. 2016 Dec 1;1(4):203-208. doi: 10.1515/pp-2016-0019. Epub 2016 Nov 25. PMID 30911624
- [Background] Graversen M, Fristrup C, Kristensen TK, Larsen TR, Pfeiffer P, Mortensen MB, Detlefsen S. Detection of free intraperitoneal tumour cells in peritoneal lavage fluid from patients with peritoneal metastasis before and after treatment with pressurised intraperitoneal aerosol chemotherapy (PIPAC). J Clin Pathol. 2019 May;72(5):368-372. doi: 10.1136/jclinpath-2018-205683. Epub 2019 Feb 12. PMID 30755498